CLINICAL TRIAL: NCT06265961
Title: Efficiency of the Bibliotherapy Method in Developing Cultural Intelligence and Competencies of Nurses: a Mixed-Methods Study
Brief Title: Efficiency of the Bibliotherapy Method in Developing Cultural Intelligence and Competencies of Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Pınar Duru, Assoc. Prof. Dr., Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 02.01.2024_39
Record Dates: First submitted 2024-02-10; First posted 2024-02-20 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Cultural Competency
MeSH Terms: interventions — Educational Status; Bibliotherapy

STUDY DESIGN:
Intervention Model Description: Mixed methods research is defined as "a research approach used in the field of health, social and behavioral sciences in which the researcher collects both quantitative and qualitative data to understand the research problems, integrates two data sets, and then draws conclusions using the advantages of integrating these two data sets." The study will be carried out in an embedded intervention research model using a combination design (Quantitative + Qualitative) in the intervention design, which is one of the advanced mixed methods designs. In the embedded mixed research model where the quantitative approach is dominant, randomized controlled research and qualitative research will be conducted simultaneously.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Education group (Active Comparator): Among the nurses who meet the inclusion criteria (N = 30), 15 nurses will be assigned to the education group after the randomization process at the beginning of the study.
  Interventions: Other: Education
- Bibliotherapy group (Active Comparator): Among the nurses who meet the inclusion criteria (N = 30), 15 nurses will be assigned to the bibliotherapy group after the randomization process at the beginning of the study.
  Interventions: Other: Education; Other: Bibliotherapy

INTERVENTIONS:
Other: Education — In line with the Papadopoulos Tilki Taylor cultural competence development model used in the research, a training presentation titled "overview and basic concepts of intercultural nursing" will be held at the beginning of the intervention in order to increase the cultural knowledge levels of nurses. In order to test the effectiveness of the bibliotherapy method, training will be given online via Google Meet to both groups (both study and control) at the beginning of the research.
Other: Bibliotherapy — The intervention consists of 1 online intercultural nursing training, 2 book and 2 short story reading activities and 1 film evaluation to be carried out over a 3-month period.
  After the training, the nurses in the study group will be asked to read the introductions of the books on the reading list and choose 2 books that they feel close to and that they have not read before. Participants will complete readings and assignments (evaluation form, reflective thought essay) asynchronously in time periods convenient to them.
  In addition to books, a supporting film will be used to raise awareness. At the end of the movie, they will be asked to write on their notes how they can relate to intercultural nursing, how they can behave when faced with similar situations, and what differences there are between their ideas about intercultural nursing before and after the movie.
  Arms: Bibliotherapy group

SUMMARY:
The study aims to evaluate the effectiveness of the developmental bibliotherapy method in developing the cultural intelligence and competence of nurses.

The study will be carried out in an embedded intervention research model using a combination design (Quantitative + Qualitative) in the intervention design, which is one of the advanced mixed methods designs. In the embedded mixed research model where the quantitative approach is dominant, randomized controlled experimental research and qualitative research will be conducted simultaneously.

1.1. Research questions for the qualitative phase 1.1.1. Research questions for the exploratory phase Q1. How successful are nurses in distinguishing the cultural differences of the individuals they care for? Q2. What are nurses' views on cross-cultural nursing care? Q4. How do nurses approach the culturally-based behaviors of the individuals they care for? Q5. What are the cultural experiences that nurses have with the individuals they care for?

1.1.2. Research questions for the integrative phase Q1. What are the contributions of the books read to the cultural intelligence and competence of nurses? Q2. What are the contributions of the stories read to the cultural intelligence and competence of nurses? Q3. What are the contributions of the watched movie to the cultural intelligence and competence of nurses?

1.1.3. Research questions for the explanatory phase Q1. What effect did bibliotherapy practice have on nurses' cultural intelligence? Q2. What impact did bibliotherapy practice have on nurses' cultural competence?

1.2. Research hypotheses of the quantitative phase

1. H1. Bibliotherapy intervention will increase the cultural intelligence levels of the nurses in the study group.
2. H1. The cultural intelligence levels of the nurses in the study group will be higher than the nurses in the control group.
3. H1. Bibliotherapy intervention will increase the cultural competence of the nurses in the study group.
4. H1. The cultural competence of the nurses in the study group will be higher than the nurses in the control group.

DETAILED DESCRIPTION:
The population of the study consists of undergraduate nurses working in Eskisehir in Türkiye. The sample of the research is; In Farokhzadian et al.'s study, cultural competence levels were reported for nursing students at the beginning (151.89±26.88) and 1 month after the intervention (184.37±22.43) in a 6-week training program implemented in a mixed design to improve cultural competence. Assuming a power of 80%, a margin of error of 0.05 and 1:1 randomization, using the values (Farokhzadian et al., 2022) as reference, it will consist of 22 nurses, 11 people in each group. Assuming that there may be losses in the study, it is planned to include 30 nurses in the study sample, with 15 people in each group, an increase of 35%.

The data collection process of the research, which will be conducted with a mixed design, will be carried out in 4 stages; In the first stage, before randomization, qualitative data will be collected by conducting in-depth interviews with all nurses included in the study through a semi-structured form for the exploratory part of the qualitative research. In the second stage, a pre-test will be applied to the study and control groups. In the third stage, data will be collected only from the study group, and will be collected in writing from the participants through a structured form for the integrative phase of the qualitative research. In the final stage, a post-test will be applied to both groups 3 months after the pre-test application, and qualitative data will be collected by conducting in-depth interviews with the nurses in the study group individually through a semi-structured form for the explanatory part of the qualitative research. The meetings will be held one-on-one via Google Meet and will be video recorded.

ELIGIBILITY:
Inclusion Criteria:

* Being a graduate nurse
* Having at least 5 years of working experience
* Working in any health institution in Eskişehir, Turkey
* Being interested and willing to read books

Exclusion Criteria:

* Not giving verbal and written consent to participate in the research.
* Working in a unit that provides outpatient treatment
* Having received post-graduate training in cross-cultural nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Cultural intelligence | From enrollment to the end of the study at 12 weeks
  In order to reveal the cultural intelligence of individuals, Ang. The "Cultural Intelligence Scale", developed by et al. in 2007 and whose Turkish validity and reliability study was conducted by İlhan and Çetin in 2017, will be used. Scale; It consists of a total of 20 items under 4 sub-dimensions named "metacognition", "cognition", "motivation" and "behavior" and has a 5-point Likert-type rating as strongly agree (5) - strongly disagree (1). The lowest score that can be obtained from the scale is 20 and the highest score is 100. High score from the scale; It means that the ability to exhibit appropriate behavior when interacting with people from different cultures, to enjoy intercultural interaction, to have self-confidence in interacting with different cultures, to acquire information about different cultures and to adjust the information acquired according to the requirements of the culture in which it interacts are developed.
Cultural competence | From enrollment to the end of the study at 12 weeks
  In order to determine the cultural competence levels of nurses, the Nurse Cultural Competence Scale, developed by Perng and Watson in 2012 and whose Turkish validity and reliability study was conducted by Gözüm et al. in 2016, will be used. Scale; It consists of a total of 20 items under 3 sub-dimensions named "cultural skill", "cultural knowledge" and "cultural sensitivity" and has a 5-point Likert type rating as strongly agree (1) - strongly disagree (5). A minimum of 20 and a maximum of 100 points can be obtained from the scale. Increasing scores from the scale indicate that the level of cultural competence has increased.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Duru, Ph.D., Principal Investigator — Eskisehir Osmangazi University
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Odunpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No